CLINICAL TRIAL: NCT00967226
Title: Propranolol vs Prednisolone for Infant Hemangiomas-A Clinical and Molecular Study
Brief Title: Propranolol Versus Prednisolone for Treatment of Symptomatic Hemangiomas
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Serious adverse events with prednisolone, primarily temporary growth retardation, <5th percentile.
Sponsor: Nancy Bauman (Other)
Responsible Party: Sponsor-Investigator, Nancy Bauman, Professor, George Washington University, Attending Children;s National, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB 4502; NIH grant number 10179326
Record Dates: First submitted 2009-08-26; First posted 2009-08-27 (Estimated); Results first posted 2016-02-24 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-01

CONDITIONS: Hemangioma of Infancy
Keywords: hemangioma
MeSH Terms: conditions — Hemangioma | interventions — Propranolol; Prednisolone; prednisolone phosphate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- propranolol for treatment of hemangiomas (Experimental): Assessing efficacy and tolerability of propranolol in management of symptomatic hemangiomas
  Interventions: Drug: propranolol
- Prednisolone (Active Comparator): Assessing efficacy and tolerability of prednisolone in management of symptomatic hemangiomas and comparing to propranolol.
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Drug: propranolol — propranolol 0.5 mg/kg orally, 4 per day - 4-6 months
  Arms: propranolol for treatment of hemangiomas
Drug: Prednisolone — 1.0 mg/kg orally, 2 per day 4-6 months
  Other Names: pediapred
  Arms: Prednisolone

SUMMARY:
Hemangiomas are relatively common lesions in infants. Most go away spontaneously after one year of life and do not need treatment. Others require treatment because they cause significant symptoms such as pain, or difficulty with breathing, eating or ambulating. Steroids have classically been used to treat hemangiomas and help to shrink them in 1/3 - 2/3 of patients. Unfortunately, steroids have many side effects in babies so physicians have sought other ways to treat them. Recently, the use of propranolol, a heart medication, was serendipitously found to reduce the size of hemangiomas. It appears to have many fewer side effects than steroids but it is not yet known if it works as well as steroids. This study seeks to compare the effect and the side effects of propranolol versus steroids for treating hemangiomas that cause symptoms in infants.

DETAILED DESCRIPTION:
Infants with symptomatic hemangiomas will be enrolled. Magnetic resonance imaging will be completed before starting medication if the extent of the hemangioma is not evident on clinical examination alone. Infants will be randomized to receive either propranolol or steroids for 4-6 months. Hemangioma response will be measured and compared monthly as will tolerability of the medications. Additionally, urine specimens will be collected at each visit to determine if markers are present that can predict response to therapy.

Additionally, any hemangiomas that are excised will be examined for genetic markers to aid in predicting response to therapy.

ELIGIBILITY:
Inclusion Criteria:

* infants with symptomatic hemangiomas

Exclusion Criteria:

* asthma
* diabetes
* hypertension
* hypotension
* hypoglycemia
* liver failure
* previous treatment for hemangiomas

Ages: 2 Weeks to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2009-07; Primary Completion 2013-01 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy M Bauman, MD, Principal Investigator — Children's Research Institute, Children's National Medical Center
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Perez RS, Mora PC, Rodriguez JD, Sanchez FR, de Torres Jde L. [Treatment of infantile hemangioma with propranolol]. An Pediatr (Barc). 2010 Feb;72(2):152-4. doi: 10.1016/j.anpedi.2009.05.019. Epub 2009 Jul 23. No abstract available. Spanish. PMID 19631595
- [Background] Denoyelle F, Leboulanger N, Enjolras O, Harris R, Roger G, Garabedian EN. Role of Propranolol in the therapeutic strategy of infantile laryngotracheal hemangioma. Int J Pediatr Otorhinolaryngol. 2009 Aug;73(8):1168-72. doi: 10.1016/j.ijporl.2009.04.025. Epub 2009 May 29. PMID 19481268
- [Background] Leaute-Labreze C, Dumas de la Roque E, Hubiche T, Boralevi F, Thambo JB, Taieb A. Propranolol for severe hemangiomas of infancy. N Engl J Med. 2008 Jun 12;358(24):2649-51. doi: 10.1056/NEJMc0708819. No abstract available. PMID 18550886
- [Derived] Bauman NM, McCarter RJ, Guzzetta PC, Shin JJ, Oh AK, Preciado DA, He J, Greene EA, Puttgen KB. Propranolol vs prednisolone for symptomatic proliferating infantile hemangiomas: a randomized clinical trial. JAMA Otolaryngol Head Neck Surg. 2014 Apr;140(4):323-30. doi: 10.1001/jamaoto.2013.6723. PMID 24526257
- [Derived] Patel NJ, Bauman NM. How should propranolol be initiated for infantile hemangiomas: inpatient versus outpatient? Laryngoscope. 2014 Jun;124(6):1279-81. doi: 10.1002/lary.24363. Epub 2013 Dec 17. No abstract available. PMID 24347141

RESULTS

PARTICIPANT FLOW:
Groups:
- Propranolol: Assessing efficacy and tolerability of propranolol in management of symptomatic hemangiomas
  propranolol: propranolol 0.67 mg/kg p.o. TID 4-6 months
- Prednisolone: Assessing efficacy and tolerability of prednisolone in management of symptomatic hemangiomas and comparing to propranolol.
  Prednisolone: 1.0 mg/kg p.o. BID 4-6 months
Period: Overall Study
Arm/Group | Propranolol | Prednisolone
Started | 11 | 8
Completed | 9 | 2
Not Completed | 2 | 6
Not completed — Adverse Event | 0 | 5
Not completed — Protocol Violation | 2 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: Infants 2 weeks - 6 months of age with symptomatic, proliferating, infantile hemangiomas
Groups:
- Propranolol: Assessing efficacy and tolerability of propranolol in management of symptomatic hemangiomas
  Propranolol 0.67 mg/kg p.o. TID x 4 - 6 months (2.0 mg/kg/day)
- Prednisolone: Assessing efficacy and tolerability of prednisolone in management of symptomatic hemangiomas and comparing to propranolol.
  Prednisolone: 1.0 mg/kg p.o. BID x 4-6 months (2.0 mg/kg/day)
- Total: Total of all reporting groups
Arm/Group | Propranolol | Prednisolone | Total
Number analyzed (Participants) | 11 | 8 | 19
Age, Continuous [Mean (Full Range); unit: months] | 4.0 [2.8 to 5.2] | 2.5 [1.7 to 3.4] | 3.4 [1.7 to 5.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 9 | 6 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 10
  Not Hispanic or Latino | 6 | 3 | 9
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 8 | 19
Total surface area (length x width) [Mean (Full Range); unit: mm squared] | 5.0 [1.9 to 25.6] | 3.1 [0.8 to 10.5] | 4.2 [0.8 to 25.6]
Adjusted total surface area (length x width x proportion of skin involved [Mean (Full Range); unit: mm squared] | 5.0 [1.5 to 24.3] | 2.5 [0.2 to 9.4] | 4.0 [0.2 to 24.3]
Ulceration [Number; unit: participants] — (not present in all participants)
  participants | 2 | 1 | 3
Morphology [Number; unit: participants] — Local, Segmental, Intermediate
  participants
    Local | 6 | 8 | 14
    Segmental | 3 | 0 | 3
    Intermediate | 2 | 0 | 2
Depth [Number; unit: participants]
  superficial | 3 | 2 | 5
  deep | 2 | 2 | 4
  mixed | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Decrease in Size of Hemangioma (Length x Width) in Square mm
Description: A priori primary outcome was proportional change in the total surface area as measured by lesion's outer margin length x width at baseline minus the same measure at 4 months with surrogate data used at 5 months if 4 months not available.
Time Frame: 4-5 months after initiating therapy
Population: Data available at 4 or 5 months for only 9/11 propranolol participants and for 6/8 prednisolone participants due to missed appointments. Overall, 90% (138/154) study appointments were completed.
Measure: Mean (95% Confidence Interval); unit: mm squared
Groups:
- Propranolol: A priori analysis, TSA (length x width) at baseline versus at 4 months with surrogate data at 5 months Propranolol 0.67 mg/kg p.o. TID x 4 - 6 months (2.0 mg/kg/day)
- Prednisolone: A priori analysis, TSA (length x width) at baseline versus at 4 months with surrogate data at 5 months
  Prednisolone: 1.0 mg/kg p.o. BID x 4-6 months (2.0 mg/kg/day)
Arm/Group | Propranolol | Prednisolone
Number analyzed (Participants) | 9 | 6
mm squared | 0.57 [0.34 to 0.80] | 0.63 [0.14 to 1.11]
Statistical Analysis 1: Comparison: Propranolol vs Prednisolone; intention to treat analysis; Test type: Superiority or Other; p = 0.77, t-test, 2 sided; Mean Difference (Net) = 0.06, Standard Deviation 0.05

2. Secondary Outcome: Tolerability of Medication
Description: All adverse events relating to medication tolerability including: adrenal crisis, growth/development, constitutional (dehydration), allergy/immunology, dermatologic, endocrine, GI, infection, metabolism/labs, pulmonary, vascular.
Time Frame: enrollment until study close out or withdrawal up to 9 months
Population: All adverse events relating to medication tolerability including: adrenal crisis, growth/development, constitutional (dehydration), allergy/immunology, dermatologic, endocrine, GI, infection, metabolism/labs, pulmonary, vascular. In this table "Adverse Events" are those exclusive of the "Serious Adverse Events" which are noted separately.
Measure: Number; unit: Events
Groups:
- Overall Number of Adverse Events in Propranolol; Overall Number of Adverse Events in Prednisolone: All (total) study adverse events displayed as "Adverse events" including mild, moderate, and severe; as well as "Serious Adverse Events"
Arm/Group | Overall Number of Adverse Events in Propranolol | Overall Number of Adverse Events in Prednisolone
Number analyzed (Participants) | 11 | 8
Events
  Adverse Events | 34 | 30
  Serious Adverse Events | 1 | 11

3. Secondary Outcome: Number of Serious Adverse Events (SAEs)
Description: Number of serious adverse events experienced by the participants in each treatment arm within the categories adrenal crisis, growth/development, constitutional. Serious adverse events are defined as events that result in death, require either inpatient hospitalization or the prolongation of hospitalization, are life-threatening, result in a persistent or significant disability/incapacity, or result in a congenital anomaly/birth defect. Other important medical events, based upon appropriate medical judgment, may also be considered Serious Adverse Events if a trial participant's health is at risk and intervention is required to prevent an outcome mentioned.
Time Frame: enrollment until study close out or withdrawal up to 9 months
Measure: Number; unit: Serious Adverse Events
Groups:
- Number of Serious Adverse Events in Propranolol: Serious adverse events in propranolol treated participants.
- Number of Serious Adverse Events in Prednisolone: Serious adverse events in prednisolone treated participants
Arm/Group | Number of Serious Adverse Events in Propranolol | Number of Serious Adverse Events in Prednisolone
Number analyzed (Participants) | 11 | 8
Serious Adverse Events | 1 | 11

4. Secondary Outcome: Growth and Development Adverse Events
Description: Number of Growth and Development AEs in each study arm
Time Frame: enrollment to study withdrawal or close out up to 9 months
Measure: Number; unit: Adverse Events
Groups:
- Growth/Developoment AEs Propranolol; Growth/Development AEs Prednisolone: Number of participants experiencing Growth/Development AEs
Arm/Group | Growth/Developoment AEs Propranolol | Growth/Development AEs Prednisolone
Number analyzed (Participants) | 11 | 8
Adverse Events | 0 | 1

5. Secondary Outcome: Pulmonary/Respiratory Adverse Events
Description: Number of pulmonary/respiratory adverse events (CTCAE 22) in each study arm
Time Frame: enrollment through study close out or withdrawal, up to 9 months
Measure: Number; unit: Adverse Events
Groups:
- Pulmonary/Respiratory AEs Propranolol; Pulmonary/Respiratory AEs Prednisolone: Number of participants experiencing pulmonary/respiratory AEs
Arm/Group | Pulmonary/Respiratory AEs Propranolol | Pulmonary/Respiratory AEs Prednisolone
Number analyzed (Participants) | 11 | 8
Adverse Events | 14 | 4

6. Secondary Outcome: Allergy/Immunology Adverse Events
Description: Number of allergy/immunology AE per study arm
Time Frame: enrollment through study closeout or study withdrawal up to 9 months
Measure: Number; unit: Adverse Events
Groups:
- Allergy/Immunology Events Propranolol: Adverse events in allergy/immunology in propranolol treated participants
- Allergy/Immunology Events Prednisolone: Adverse events in allergy/immunology in prednisolone treated participants
Arm/Group | Allergy/Immunology Events Propranolol | Allergy/Immunology Events Prednisolone
Number analyzed (Participants) | 11 | 8
Adverse Events | 1 | 1

7. Secondary Outcome: Dermatologic Adverse Events
Description: Number of Dermatologic Adverse Events in each study arm.
Time Frame: enrollment to study close out or withdrawal up to 9 months
Measure: Number; unit: Adverse Events
Groups:
- Dermatologic AEs Propranolol; Dermatologic AEs Prednisolone: Number of participants experiencing Dermatologic AEs
Arm/Group | Dermatologic AEs Propranolol | Dermatologic AEs Prednisolone
Number analyzed (Participants) | 11 | 8
Adverse Events | 2 | 1

8. Secondary Outcome: Endocrinologic Adverse Events
Description: Number of Endocrinologic AEs (of which adrenal crisis does not overlap).
Time Frame: enrollment to close out or study withdrawal up to 9 months
Measure: Number; unit: Adverse Events
Groups:
- Endocrine AEs Propranolol; Endocrinologic AEs Prednisolone: Number of participants experiencing Endocrinologic AEs.
Arm/Group | Endocrine AEs Propranolol | Endocrinologic AEs Prednisolone
Number analyzed (Participants) | 11 | 8
Adverse Events | 0 | 7

9. Secondary Outcome: Gastrointestinal Adverse Events
Description: Number of Gastrointestinal AEs in each arm
Time Frame: enrollment to study withdrawal or study close out up to 9 months
Measure: Number; unit: Adverse Events
Groups:
- Gastrointestinal AEs Propranolol; Gastrointestinal AEs Prednisolone: Number of Participants experiencing Gastrointestinal AEs
Arm/Group | Gastrointestinal AEs Propranolol | Gastrointestinal AEs Prednisolone
Number analyzed (Participants) | 11 | 8
Adverse Events | 6 | 6

10. Secondary Outcome: Infectious Adverse Events
Description: Number of infectious AEs in each study arm (i.e. conjunctivitis, thrush, fever)
Time Frame: enrollment to study withdrawal or close out up to 9 months
Measure: Number; unit: Adverse Events
Groups:
- Infectious AEs Propranolol; Infectious AEs Prednisolone: Number of participants experiencing Infectious AEs
Arm/Group | Infectious AEs Propranolol | Infectious AEs Prednisolone
Number analyzed (Participants) | 11 | 8
Adverse Events | 5 | 3

11. Secondary Outcome: Metabolic or Laboratory AEs
Description: Number of Metabolic or Laboratory AEs in each study arm.
Time Frame: enrollment to study withdrawal or close out up to 9 months
Measure: Number; unit: Adverse Events
Groups:
- Metabolic/Laboratory AEs Propranolol: Number of participants experiencing Metabolic or Laboratory AEs.
- Metabolic/Laboratory AEs Prednisolone: Number of participants experiencing Metabolic or Laboratory AEs in each study arm.
Arm/Group | Metabolic/Laboratory AEs Propranolol | Metabolic/Laboratory AEs Prednisolone
Number analyzed (Participants) | 11 | 8
Adverse Events | 1 | 0

12. Secondary Outcome: Vascular Adverse Events
Description: Number of Vascular AEs in each study arm.
Time Frame: enrollment to study withdrawal or close out up to 9 months
Measure: Number; unit: Adverse Events
Groups:
- Vascular AEs Propranolol; Vascular AEs Prednisolone: Number of participants experiencing Vascular AEs
Arm/Group | Vascular AEs Propranolol | Vascular AEs Prednisolone
Number analyzed (Participants) | 11 | 8
Adverse Events | 3 | 4

13. Secondary Outcome: Constitutional Adverse Events
Description: Number of constitutional AEs in each study arm.
Time Frame: enrollment to study close out or withdrawal up to 9 months
Measure: Number; unit: Adverse Events
Groups:
- Constitutional AEs Propranolol; Constitutional AEs Prednisolone: Number of Participants experiencing Constitutional AEs
Arm/Group | Constitutional AEs Propranolol | Constitutional AEs Prednisolone
Number analyzed (Participants) | 11 | 8
Adverse Events | 2 | 3

ADVERSE EVENTS:
Time Frame: Adverse events collected in first 9 months participants treated with medication.
Groups:
- Propranolol: Assessing efficacy and tolerability of propranolol in management of symptomatic hemangiomas
  propranolol: propranolol 0.5 mg/kg p.o. QID 6 months or less
- Prednisolone: Assessing efficacy and tolerability of prednisolone in management of symptomatic hemangiomas and comparing to propranolol.
  Prednisolone: 1.0 mg/kg p.o. BID x 6 months or less
Arm/Group | Propranolol | Prednisolone
Serious Adverse Events (participants affected / at risk) | 1/11 | 5/8
Other Adverse Events (participants affected / at risk) | 11/11 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Propranolol (N=11) | Prednisolone (N=8)
Adrenal Crisis (Endocrine disorders) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 5 (9)
Dehydration (General disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Propranolol (N=11) | Prednisolone (N=8)
Dermatologic (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Gastrointerstinal (Gastrointestinal disorders) | 5 (6) | 5 (6)
Infection (Infections and infestations) | 2 (5) | 2 (3)
Metabolic/Lab (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pulmonary/respiratory (Respiratory, thoracic and mediastinal disorders) | 8 (14) | 3 (4)
Vascular (Vascular disorders) | 3 (3) | 1 (4)
Endo (Endocrine disorders) | 0 (0) | 6 (7)
Allergy (General disorders) | 1 (1) | 1 (1)
Constitutional (General disorders) | 2 (2) | 3 (3)
Growth suppression (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Not every enrolled participant had an adverse event and some had more than one. The prednioslone participants who had adverse events warranting early withdrawal had severe failure to thrive (<5th percentile), a serious adverse event.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No